CLINICAL TRIAL: NCT04733690
Title: METABOLIC (GLYCEMIC, INSULINEMIC & SATIETY) CHARACTERISTICS OF A NOVEL COMMON BEAN (Phaseolus Vulgaris L.) PRODUCT
Brief Title: METABOLIC CHARACTERISTICS OF A NOVEL COMMON BEAN PRODUCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jomo Kenyatta University of Agriculture and Technology (Other)
Collaborators: KU Leuven (Other); Legumes Centre of Excellence for Food and Nutrition Security (Unknown); VLIR-UOS (Unknown)
Responsible Party: Principal Investigator, Dr. Florence Kyallo, Senor Lecturer, Jomo Kenyatta University of Agriculture and Technology
Other Study IDs: P751-2020
Record Dates: First submitted 2021-01-27; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes
Keywords: Phaseolus vulgaris L.; Glycemic Index; Food Insulin Index; Appetite; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteers (Glycemic Index): The glycemic index (GI) of the common bean product will be assessed in this cohort among 10 study participants. The GI of the product will be assessed on 3 test days over a 120 min period on each study day.
  Interventions: Dietary Supplement: Common bean product
- Healthy Volunteers(Food Insulin Index): The food insulin index (FII) of the common bean product will be assessed in this cohort among 10 study participants. This study will recruit 10 participants. The FII of the product will be assessed on 3 test days over a 120 min period on each study day.
  Interventions: Dietary Supplement: Common bean product
- Type-2 diabetes (T2DM) patients: Glycemic, insulinemic and satiety responses associated with the consumption of the common bean product will be assessed in this cohort among 10 T2DM patients. Participants will attend one study visit lasting approximately 120 min.
  Interventions: Dietary Supplement: Common bean product

INTERVENTIONS:
Dietary Supplement: Common bean product — Healthy volunteers Healthy volunteers in the GI and FII studies will participate in the study during 3 test days for each of the studies. The reference food will be tested 2 times and the test food 1 time in each participant.
  T2DM patients T2DM patients will participate in the study for one test day for the assessment of postprandial glycemic, insulinemic and satiety responses.
  For both healthy volunteers and T2DM patients, the following will be assessed during study days: 24-hour of dietary recall; weight, height, waist and hip circumferences; blood pressure; and body composition using bioelectrical impedance analysis (BIA). Participants will be fed with a portion of the test or reference food and 250ml water. Two fasting blood samples (-5 and 0 min) and postprandial blood samples (15, 30, 45, 60, 90 and 120 min) will be collected

SUMMARY:
Kenya is classified as having three main forms of malnutrition (overweight, anaemia and stunting), exhibiting a double burden of malnutrition nutritional landscape. Trends from the 80s to present show that indicators of overweight and obesity, and diabetes in both adult men and women either show no progress or are worsening. It is a chronic inflammatory metabolic disease occurring when the pancreas is unable to produce sufficient amounts of insulin or when the body cannot effectively utilize produced insulin or both.

Given that T2DM impacts on several aspects of a patient's quality of life, functionality, and health status, finding effective dietary strategies to combat this condition is key. In diabetes patients, low-glycemic index foods rich in dietary fibre, vitamins, and minerals should be encouraged. Common beans are an important source of iron and zinc. Common beans contain slowly digestible carbohydrates and a high proportion of non-digestible carbohydrates. Fibre (soluble and non-soluble) in beans would be beneficial to T2DM patients by reducing macronutrient absorption, satiety increase, increased sensibility to insulin, effects on inflammatory markers and on intestinal microbiota. Moreover, they contain several bioactive compounds possessing anti-inflammatory, antioxidant and other biological activity. Due to their composition and effects, common beans have attractive properties for T2DM patients. The common bean predominates other legumes in terms of production in Africa. The aim of this research is to study the associated glucose, insulin and appetite responses associated with the consumption of a novel common bean product.

DETAILED DESCRIPTION:
Type-2 diabetes (T2DM) in Kenya is on a rise with about 458,900 people diagnosed in 2017 and a 2.5-fold projected increase by 2030. Prevalence of T2DM is 5.8% and 6.2% in men and women. T2DM has an inflammatory disease character and is characterized by hyperglycemia. Common beans in T2DM patients could have many health benefits such as modulation of glucose metabolism, reduction of low-density lipoproteins, and satiety.

In this research, we develop a food-grade novel common bean product from food-grade ingredients though the application of conventional food processing technologies. We will then assess postprandial insulin, blood glucose and appetite responses associated with consumption of the common bean product in healthy volunteers and T2DM patients. The specific aims of our research are:

1. to assess the glycemic index (GI) of the common bean product in vivo among 10 healthy volunteers. The GI of the product will be measured over a 120 min period starting at the ingestion of the common bean product. Participants will be fed with an equi-carbohydrate portion of the common bean product to the reference food (anhydrous glucose powder, 50g or dextrose (glucose monohydrate), 55g). The test food and reference food will be assessed in each subject on separate days with a 1 week period between each study day.
2. to assess the food insulin index (FII) of the common bean product in vivo among 10 healthy volunteers. Participants will be fed with iso-caloric (240 kilocalorie) portions of the test food and reference food.
3. to determine glycemic, insulinemic and satiety (appetite) response associated with consumption of the common bean product among T2DM patients. Glycemic and insulinemic response will be evaluated over a 120 min period starting at the ingestion of the common bean product. Appetite scores will be used to assess the satiety power of the test product. The appetite score will be assessed before and after consumption of test product at time points 0, 15, 30, 45, 60, 90 and 120 minutes using short questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (incl. criteria)

  * Male or female 18-69 years
  * No known food allergies or intolerances
  * No prescription medication (excluding oral contraceptives) known to affect glucose intolerance (e.g. steroids, protease inhibitors, antipsychotics e.t.c.)
* T2DM patients (incl. criteria)

  * Male or female aged 18-69 years
  * Previously diagnosed with type 2 diabetes
  * Consenting to participate

Exclusion Criteria:

* Healthy volunteers (excl. criteria)

  * Known history of diabetes mellitus or use of anti-hyperglycaemic medication or insulin
  * Alcohol or tobacco use in the evening preceding the test
  * Vigorous exercise on the morning of the test
  * Undergone major medical/surgical event needing hospitalization within the preceding 3 months
  * Presence of disease or drug influencing digestion and absorption of medicine
* T2DM patients (excl. criteria)

  * Use of prescription medication
  * History of eating disorders and irregular eating habits
  * Use of tobacco or alcohol
  * Females experiencing menstrual period or adverse premenstrual symptoms

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers The healthy volunteers will be recruited from Jomo Kenyatta University of Agriculture and Technology (JKUAT) and handled at the JKUAT University Hospital.
  T2DM patients The participants will be recruited from the Makueni Level-5 and Mbooni sub-county hospitals which run a diabetes outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-02-04 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic response | 120 min
  The effect associated with consumption of the common bean product on blood sugar (glucose) levels.
Insulinemic response | 120 min
  The effect associated with consumption of the common bean product on insulin levels.
Satiety | 120 min
  Appetite score refers to the average between hunger, desire to eat, prospective consumption and a 100-fullness score.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be stored by the principal investigators. A controlled access approach, allowing for review of requests will be used to provide secure data access. Study findings will be published in peer-reviewed journals and also presented in conferences, research seminars and workshops through oral or poster presentations after completion of this study.

REFERENCES:
- [Background] ISO, "ISO 26642:2010(en), Food products - Determination of the glycaemic index (GI) and recommendation for food classification," 2010. [Online]. Available: https://www.iso.org/obp/ui/#iso:std:iso:26642:ed-1:v1:en. [Accessed: 04-Jul-2019].

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-31): https://cdn.clinicaltrials.gov/large-docs/90/NCT04733690/Prot_SAP_ICF_000.pdf